CLINICAL TRIAL: NCT06774911
Title: Evaluation of Amino Acids Bioavailability in a Food Product Based on a Vegetable Protein Combination: A Randomized, Double-blind Crossover Study
Brief Title: Evaluation of Amino Acids Bioavailability in a Food Product Based on a Vegetable Protein Combination
Acronym: BIODISPROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: ANFACO-CECOPESCA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BIODISPROT
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Biological Availability; Bioavailability and AUC
Keywords: vegetal proteins; Inflammation; Satiety; Hunger; Amino acids
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Crossover, Randomized, Double-Blind Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protein from rice and pea (YUIT) (Experimental): Participants will receive 100g of powdered product with a complete and balanced nutritional profile with pea and rice protein source + 500 mL of water.
  Interventions: Other: YUIT
- Protein from soy (P_PS) (Active Comparator): Participants will receive 94.5 g of powdered product with a complete and balanced nutritional profile (the same as the YUIT product) with soy protein source + 500 mL of water
  Interventions: Other: P_PS

INTERVENTIONS:
Other: YUIT — Product with protein source from pea and rice.
  Arms: Protein from rice and pea (YUIT)
Other: P_PS — Product with protein source from soy protein.
  Arms: Protein from soy (P_PS)

SUMMARY:
Proteins can be classified as high or low biological value proteins depending on their composition in essential amino acids, which are those amino acids that the body cannot synthesize and must be provided through food. In recent years, there has been growing interest in reducing the consumption of proteins of animal origin, leading to the search for more sustainable protein options, such as vegetable proteins. However, vegetable options do not have a complete profile of essential amino acids. In this sense, soy protein is considered the reference vegetable protein because it has an adequate amino acid profile. However, the amount of methionine is considerably lower than that of an animal source, and it also has a considerable allergenic potential. The mixture of two types of complementary vegetable protein sources could serve as a strategy to achieve the profile of essential amino acids like that of an animal protein.

The hypothesis of the present study is that the consumption of a mixture of vegetable proteins from legume and cereal sources will complement each other to achieve a bioavailability of essential amino acids equal to or greater than that observed when consuming soy protein.

DETAILED DESCRIPTION:
An adequate protein intake is essential for the body's well-being and performance, because the body uses this nutrient in many cellular functions.

Proteins are nitrogen-containing substances made up of amino acids (AA). Not only the quantity but also the quality of protein in the diet is important for the body's proper functioning. Protein quality depends on the AA profile, among other factors. 20 total AA (TAA) have been identified as necessary for human growth and metabolism. Of the 20 TAAs, nine of them are defined as essential AA (EAAs, histidine, isoleucine, leucine, lysine, methionine, phenylalanine, threonine, tryptophan and valine), and the remaining eleven are considered non-essential AA (NEAAs, alanine, arginine, asparagine, aspartic acid, cysteine, glutamic acid, glutamine, glycine, proline, serine and tyrosine). In addition, branched-chain amino acids (BCAA, leucine, isoleucine, and valine) are found within the EAAs.

The NEAAs can be synthesized by the body, while the EAAs must be ingested from the diet. In this sense, proteins can be classified into two groups: high or low biological value, depending on the presence or absence of all the EAAs in their composition. Today, this distinction is usually called animal or vegetable proteins, respectively, because proteins from meat, eggs, and dairy products have higher amounts of EAAs, including leucine, while proteins from legumes, seeds, or nuts have a deficit in some of them.

In the diet, the consumption of a mixture of plant-based proteins (i.e., complementary proteins) is a common strategy to compensate for the fact that individual sources of plant-based proteins are often deficient in one or more EAAs. For example, the combination of rice protein (high in methionine but low in lysine) and pea protein (low in methionine but high in lysine) can produce a pea-rice protein blend with a balanced amino acid profile, free of deficiencies. Therefore, the formulation of a plant-based protein blend represents an opportunity to develop a high-quality protein option.

The present study has as its main objective to evaluate the postprandial bioavailability of EAA from two plant-based protein sources present in a complete powdered meal, where one will have soy protein and the other product with a protein source from a mixture of rice and pea protein.

The secondary objectives of the study are to compare the following kinetic parameters and the metabolic response of the two products with different plant-based protein sources.

* Bioavailability of AAT (AAT-AUC0-240min), AANE (AANE-AUC0-240min), BCAA (BCAA-AUC0-240min) and of each of the EAA individually (EAA-AUC0-240min).
* Time to reach maximum concentration of AAT (AAT-Tmax), AAE (AAE-Tmax), AANE (AANE-Tmax), BCAA (BCAA-Tmax) and of each EAA individually.
* Maximum concentration of AAT (AAT-CMax), AAE (AAE-CMax), AANE (AANE-CMax), BCAA (BCAA-CMax) and of each EAA individually.
* Insulinotropic response: insulin and blood glucose levels.
* Objective hunger and satiety modulation: blood levels of hunger and satiety regulating hormones: glucagon-like peptide-1 (GLP-1), peptide YY (PPY), ghrelin.
* Modulation of hunger and subjective satiety.
* Changes in the expression of genes involved in oxidative and inflammatory metabolism.

During the study there will be 3 visits: a preselection visit (V0), a visit for the first postprandial study (V1) and after one week washing period, a visit for the second postprandial study (V2).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 50 years old.
* Be willing to limit intentional physical exercise during the 24 hours prior to each day of testing.
* Be willing to not consume alcoholic beverages 48 hours before the start of the study.
* Sign the informed consent.
* Be able to read, write and speak Spanish.

Exclusion Criteria:

* Present values of body mass index (BMI) ≤ 18kg/m^2 or ≥ 30 kg/m^2.
* Present allergy or intolerance to any of the ingredients of the products to be evaluated, mainly pea flour, rice flour, soy, flax, spirulina or olive oil.
* Follow a vegan or vegetarian diet.
* Use of medication that affects muscle anabolism or metabolism in general.
* Consume multivitamin supplements (Vit. D, Vit. E and Vit. C), minerals (Zinc, Selenium), essential fatty acids (omega-3), polyphenols, or any type of supplements that may affect oxidative or inflammatory metabolic pathways in the last 30 days before the start of the study.
* Consumption of alcoholic beverages:

  * Men: consume 4 or more Standard Drink Units (SDU) daily or 28 SDU weekly.
  * Women: Consume 2 or more Standard Drink Units (SDU) daily or 17 SDU weekly.
* Be an active smoker or have been one less than 6 months ago.
* Have a chronic disease with clinical manifestations: coronary disease, cardiovascular disease, diabetes, celiac disease, Crohn's disease, chronic kidney disease, active cancer, gastrointestinal diseases that may compromise the absorption of the compound.
* Take protein or amino acid supplements up to 1 week before the start of the study.
* Perform vigorous exercise for more than 3 hours a week.
* Have anemia.
* Have lost 3 kg or more in the last 3 months.
* Be pregnant or intend to become pregnant.
* Be breastfeeding.
* Not be able to follow the study guidelines.
* Be participating or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Bioavailability of essential aminoacids calculated by the Area Under The Curve (EAA-AUC 0-240min) of plasma essential aminoacids levels. | At week 1 and week 2
  Fasting EAA levels in plasma will be determined before consuming the products until 4 hours postprandially at 6 points after consuming the product (30 min., 60min., 90min., 120 min., 180 min., 240 min.).
  Plasma EAA will be quantified by liquid chromatography coupled to triple quadrupole mass spectrometry (LC-MS/MS).

SECONDARY OUTCOMES:
Bioavailability of total amino acids (TAA-AUC0-240 min) levels in plasma. | At week 1 and week 2
  Fasting TAA levels in plasma will be determined before consuming the product until 4 hours postprandially at 6 points after consuming the product ( 30 min., 60min., 90 min., 120 min., 180 min., 240 min.).
  Plasma TAA will be quantified by liquid chromatography coupled to triple quadrupole mass spectrometry (LC-MS/MS).
Bioavailability of non-essential amino acids (NEAA-AUC0-240 min) levels in plasma. | At week 1 and week 2
  Fasting NEAA levels in plasma will be determined before consuming the product until 4 hours postprandially at 6 points after consuming the product (30 min., 60min., 90 min., 120 min., 180 min., 240 min.).
  Plasma NEAA will be quantified by liquid chromatography coupled to triple quadrupole mass spectrometry (LC-MS/MS).
Bioavailability of branched chain amino acids (BCAA-AUC0-240min) levels in plasma. | At week 1 and week 2
  Fasting BCAA levels in plasma will be determined before consuming the product until 4 hours postprandially at 6 points after consuming the product ( 30 min., 60min., 90 min., 120 min., 180 min., 240 min.).
  Plasma BCAA will be quantified by liquid chromatography coupled to triple quadrupole mass spectrometry (LC-MS/MS).
Bioavailability of each of the essential amino acids individually (AUC0-240min) levels in plasma. | At week 1 and week 2
  Fasting each essential aminoacids levels in plasma will be determined before consuming the product until 4 hours postprandially at 6 points after consuming the product ( 30 min., 60min., 90 min., 120 min., 180 min., 240 min.).
  Plasma each essential aminoacids levels will be quantified by liquid chromatography coupled to triple quadrupole mass spectrometry (LC-MS/MS).
Time for maximum plasma concentration (Tmax) | At week 1 and week 2
  Time period for the maximum plasma concentration of TAA, NEAA, BCAA and each essential aminoacids
Maximum plasma concentration (Cmax) | At week 1 and week 2
  Maximum plasma concentration of TAA, NEAA, BCAA and each essential aminoacids.
Insulinotropic response: Change in serum insulin levels (mU/L). | At week 1 and week 2
  Fasting insulin levels in serum will be determined before consuming the product until 3 hours postprandially at 7 points after consuming the product (15min., 30min., 45min., 60min., 90min., 120min. and 180min.) Insulin levels will be measured by standardized chemiluminescence methods.
Insulinotropic response: Change in serum glucose levels (mg/dL). | At week 1 and week 2
  Fasting glucose levels in serum will be determined before consuming the product until 3 hours postprandially at 7 points after consuming the product (15min., 30min., 45min., 60min., 90min., 120min. and 180min.) Serum glucose levels will be determined by standardized spectrophotometry methods.
Change of blood glucagon-like peptide-1 (GLP-1) levels (ng/mL). | At week 1 and week 2
  Levels of blood GLP-1, will be measured by standardized chemiluminescence methods at extraction points: 0min., 30min., 60min., 120min., 180min. and 240 min.
Change of blood peptide YY (PPY) levels (pg/mL). | At week 1 and week 2
  Levels of blood PPY, will be measured by standardized chemiluminescence methods at extraction points: 0min., 30min., 60min., 120min., 180min. and 240 min.
Change of blood ghrelin levels (pg/mL) | At week 1 and week 2
  Levels of blood ghrelin will be measured by standardized chemiluminescence methods at extraction points: 0min., 30min., 60min., 120min., 180min. and 240 min.
Modulation of subjective hunger | At week 1 and week 2
  The evaluation of the sensation of subjective hunger will be assessed by using a 100 mm Visual Analogue Scale (VAS) at the following points: 0 min (baseline time), 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 180 and 240 min.
  The VAS is presented as a horizontal line 100 mm long, with two ends that represent the limits of the phenomenon to be evaluated: One end of the line is labeled "No hunger" (0), while the other end is marked as "extreme hunger" (100). The volunteer is asked to mark on the line the point that best represents the intensity of what he or she is feeling at that moment. The mark made is measured in millimeters from the bottom end (zero), and the value obtained is the quantitative representation of the phenomenon evaluated.
Modulation of subjective satiety | At week 1 and week 2
  The evaluation of the sensation of subjective satiety will be assessed by using a 100 mm Visual Analogue Scale (VAS) at the following points: 0 min (baseline time), 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 180 and 240 min.
  The VAS is presented as a horizontal line 100 mm long, with two ends that represent the limits of the phenomenon to be evaluated: One end of the line is labeled "not at all satisfied" (0), while the other end is marked as "totally satisfied" (100). The volunteer is asked to mark on the line the point that best represents the intensity of what he or she is feeling at that moment. The mark made is measured in millimeters from the bottom end (zero), and the value obtained is the quantitative representation of the phenomenon evaluated.
Modulation of subjective fullness. | At week 1 and week 2
  The evaluation of the sensation of subjective fullnes will be assessed by using a 100 mm Visual Analogue Scale (VAS) at the following points: 0 min (baseline time), 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 180 and 240 min.
  The VAS is presented as a horizontal line 100 mm long, with two ends that represent the limits of the phenomenon to be evaluated: One end of the line is labeled "no feeling of fullness" (0), while the other end is marked as "I have the greatest feeling of fullness I have ever had" (100). The volunteer is asked to mark on the line the point that best represents the intensity of what he or she is feeling at that moment. The mark made is measured in millimeters from the bottom end (zero), and the value obtained is the quantitative representation of the phenomenon evaluated.
Modulation of subjective desire to eat food. | At week 1 and week 2
  The evaluation of the sensation of subjective fullnes will be assessed by using a 100 mm Visual Analogue Scale (VAS) at the following points: 0 min (baseline time), 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 180 and 240 min.
  The VAS is presented as a horizontal line 100 mm long, with two ends that represent the limits of the phenomenon to be evaluated: One end of the line is labeled "I have no desire to eat food" (0), while the other end is marked as "I have the greatest desire to eat any food" (100). The volunteer is asked to mark on the line the point that best represents the intensity of what he or she is feeling at that moment. The mark made is measured in millimeters from the bottom end (zero), and the value obtained is the quantitative representation of the phenomenon evaluated.
Modulation of subjective desire to eat anything fatty, salty, sweet or tasty. | At week 1 and week 2
  The evaluation of the sensation of subjective desire to eat anything fatty, salty, sweet or tasty.will be assessed by using a 100 mm Visual Analogue Scale (VAS) at the following points: 0 min (baseline time), 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 180 and 240 min.
  The VAS is presented as a horizontal line 100 mm long, with two ends that represent the limits of the phenomenon to be evaluated: One end of the line is labeled "I have no desire to eat anything fatty, salty, sweet or tasty" (0), while the other end is marked as "I have the greatest desire to eat anything fatty, salty, sweet or tasty" (100). The volunteer is asked to mark on the line the point that best represents the intensity of what he or she is feeling at that moment. The mark made is measured in millimeters from the bottom end (zero), and the value obtained is the quantitative representation of the phenomenon evaluated.
Expression of genes involved in inflammatory and oxidative metabolism | At week 1 and week 2
  Changes in gene expression of genes involved in oxidative and inflammatory pathways will be quantified by transcriptomics of blood samples at baseline and at 240 min.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari PhD, Principal Investigator — Fundació Eurecat
Locations (1):
- Eurecat, Reus, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org